CLINICAL TRIAL: NCT04711538
Title: Role of Diagnostic Imaging in Evaluation of Cochlear Implant Candidate
Brief Title: Role of Diagnostic Imaging in Cochlear Implant
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Marwa Helmy Abdel Hamid Elhadad, doctor, Sohag University
Other Study IDs: Soh-Med-21-01-05
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Cochlear Implant
MeSH Terms: interventions — Postmortem Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MRI — imaging inner ear and petrous bone of the candidate by MRI and CT
  Other Names: CT imaging

SUMMARY:
cochlear implant is a well accepted treatment to profound sensorineural hearing loss. Imaging provides essential information about anatomical Variants that could be riskyand should be considered by cochlear implant surgeon and the aim of the study:-

* Identify inner ear congenital and acquired abnormalities.
* Identify cochlear nerve anomalies.
* Detect temporal bone abnormalities that require surgical modification by cochlear implant surgeon.

DETAILED DESCRIPTION:
Cochlear implant (CI) is a well-accepted treatment for severe to profound sensorineural hearing loss. Patients who are refractory to conventional hearing augmentation .

(CI) is a surgically implanted device consisting of external and internal components. An external microphone and speech processor worn behind the ear and convert sound into an electrical signal. A magnet held external transmitter sends the signal via electromagnetic induction through the skin to an internal receiver- stimulator which converts the signal into rapid electrical impulses which distributed to multiple electrodes on an electrode array implanted within the cochlea. The electrodes electrically stimulate the spiral ganglion cells along the cochlear turns, which then travel along the auditory nerve axons to the brain for sound perception .

Imaging provides essential information about many of the anatomical variations that could be risky and should be considered by cochlear implant surgeon to avoid complications.

Some variations are potential surgical hazards that may lead to problems during the surgery and may alert the surgeon regarding potential surgical dangers and complications .

Both computed tomography (CT) and magnetic resonance imaging(MRI) are complementary to each other. They detect cochlear, middle ear anatomy and the anatomical variants .

The strength of CT is visualization of the bony structures of the middle and inner ear and the strength of MRI is visualization of the fluid content of the membranous labyrinth, visualization of the vestibule-cochlear nerve in the fluid filled internal auditory canal and the cerebello-pontine angle .

ELIGIBILITY:
Inclusion Criteria:

* Age, any age will included
* Gender, both genders will be included.
* Patient full filled criteria for CI including audiological & phoniatric criteria

Exclusion Criteria:

* • Patient who did not fulfill the criteria for indicating CI surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients who suffering from deep to profound sensorineural hearing loss( inculde any age,both genders)
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
identification inner ear congenital and acquired abnormalities | immediately after end of imaging and diagnosis
  detect role of MRI and CT in identification of cochlear nerve anomlies,detect temporal bone abnormalities that require surgical modification by cochlear implant surgeon.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed H Alam-Eldeen, AP, Study Director — Sohag University; Ramadan H Hashem, Prof, Study Chair — Sohag University
Locations (1):
- Sohag University, Sohag, Sohag Governorate, Egypt

REFERENCES:
- [Background] Alam-Eldeen MH, Rashad UM, Ali AHA. Radiological requirements for surgical planning in cochlear implant candidates. Indian J Radiol Imaging. 2017 Jul-Sep;27(3):274-281. doi: 10.4103/ijri.IJRI_55_17. PMID 29089672
- [Result] Joshi VM, Navlekar SK, Kishore GR, Reddy KJ, Kumar EC. CT and MR imaging of the inner ear and brain in children with congenital sensorineural hearing loss. Radiographics. 2012 May-Jun;32(3):683-98. doi: 10.1148/rg.323115073. PMID 22582354
- [Result] Marsot-Dupuch K, Meyer B. Cochlear implant assessment: imaging issues. Eur J Radiol. 2001 Nov;40(2):119-32. doi: 10.1016/s0720-048x(01)00380-1. PMID 11704359